CLINICAL TRIAL: NCT03679845
Title: A Pilot Study to Assess the Safety and Efficacy of Sarilumab in Halting Progression of Morphea
Brief Title: Study to Assess Sarilumab in Halting Progression of Morphea
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Difficulty in recruiting patients
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Gideon Piers Smith, Medical Director Department of Dermatology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018P002128
Record Dates: First submitted 2018-09-17; First posted 2018-09-20 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Morphea, Plaque Form
MeSH Terms: conditions — Scleroderma, Localized | interventions — sarilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Sarilumab Arm (Experimental): 200 mg of sarilumab every two weeks
  Interventions: Drug: Sarilumab

INTERVENTIONS:
Drug: Sarilumab — Sarilumab is an IL-6 monoclonal antibody that has shown to be potentially important in the creation of sclerosis in SSc.
  Other Names: Kevzara

SUMMARY:
An open-label single center trial studying the efficacy and safety of sarilumab on morphea patients.

DETAILED DESCRIPTION:
Morphea, like systemic sclerosis (SSc), presents with sclerotic hardening of the skin. However, unlike SSc, morphea has no systemic involvement. While this skin-limited, chronic sclerosis, has no impact on mortality, it can have significant morbidity, as lesions can affect joint mobility, and be disfiguring, especially when involving the face. While some patients respond well to use of steroids, whether topical or intralesional, antimalarials such as plaquenil, or traditional immuno-suppressants there is a significant proportion of patients who remain non-responsive to these treatments, or require high dosages of these, oral steroids, or experimental therapies to suppress the condition. For this group of patients there is a high clinical need to find alternate therapies. In addition, as the disease creates permanent scarring, and traditional immuno-suppressants take several months to take effect there is a need for medications that can act more quickly to halt the progression of scarring.

Although the pathways of inflammation are poorly understood, one cytokine of potential interest is IL (interleukin)-6. In the bleomycin mouse model of skin sclerosis targeting IL-6 by both passive and active immunization strategies prevented the development of bleomycin-induced dermal fibrosis. Dysregulation of IL-6 has also been seen in the serum of patients suffering from SSc. As a result, preliminary clinical trials have been undertaken in SSc. While results did not reach statistical significance the skin thickening was better in the treatment group than in placebo and the lack of signal is likely due to the late stage of patients skin involvement, and the slow progression of thickening in SSc. In contrast morphea often progresses rapidly and as such is much more likely to give a clear clinical signal.

Recently sarilumab, an anti-IL-6 monoclonal antibody, has been approved for use in severe rheumatoid arthritis (RA) after rapid and sustained results in clinical trials. Given its good safety profile, its impressive response in RA, and the immunohistochemical evidence that IL-6 may be important in creation of sclerosis in SSc, the investigators propose a pilot study to determine the safety and efficacy of sarilumab in morphea.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject 18 years of age or older
2. Only circumscribed (plaque) morphea with at least one active morphea target lesion (0.5-10 cm2), with mLoSSI ≥ 5.
3. Body surface area affected by morphea lesions: ≤ 50% at start of treatment
4. If subject has received any morphea treatment, subject must be on a stable regimen, which is defined as not starting a new drug or changing dosage within 8 weeks prior to Day 1. Subject must be willing to stay on a stable regimen during the duration of the study.
5. Willingness of subject to follow all study procedures
6. Willingness to avoid excessive exposure of diseased areas to natural or artificial sunlight

Exclusion Criteria:

1. Use any topical medication treating morphea within 14 days prior to Day 1
2. Pregnancy or breast feeding
3. Any condition (e.g. HIV, diabetes, ANC(absolute neutrophil count) < 2,000/mm3, platelets < 150,000/mm3 or AST(aspartate transaminase)/ALT(alanine aminotransferase) > 1.5 times normal limits) or therapy that in the investigator's opinion may pose a risk to the subject or that could interfere with any evaluation in the study
4. Cancer within 5 years other than non-melanoma skin cancer or cervical cancer in situ that has been fully treated.
5. Known hypersensitivity to any of the constituents or excipients of the investigational product
6. Use of any prescription or non-prescription medication that could interfere with efficacy evaluations in the study
7. Participation in another clinical research study with an investigational drug within 4 weeks before this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
efficacy of sarilumab in plaque type morphea | Week 24
  To determine the efficacy of sarilumab in plaque type morphea by clinical responder rate at week 24.

SECONDARY OUTCOMES:
Physician Global Assessment of Activity (PGA-A) | Baseline and Week 24
  100-mm morphea activity scale anchored by "inactive" at 0 and "markedly active" at 100.

CONTACTS AND LOCATIONS:
Locations (1):
- CURTIS (Massachusetts General Hospital), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No